CLINICAL TRIAL: NCT04859361
Title: Comparison of Conservative Treatment of Cervical Intraepithelial Lesions With Imiquimod With Standard Excisional Technique Using LLETZ: a Randomized Controlled Trial
Brief Title: Comparison of Treatment of Cervical Intraepithelial Lesions With Imiquimod or LLETZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01-02
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Intraepithelial Neoplasia, Cervical
Keywords: imiquimod; LLETZ; cervical intraepithelial lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with imiquimod (Experimental): Colposcopy with PAP smear and punch biopsy is scheduled at 10 weeks to rule out progression, and at 20 weeks to evaluate treatment success. At 20 weeks, biopsies will be performed at the locations where lesions were previously present and additional biopsies will be performed on any visible lesions. At 20 weeks, in case of disease progression or persistence, treatment with LLETZ will be offered.
  Interventions: Drug: Aldara 5% Topical Cream
- Treatment with LLETZ (Active Comparator): Standard treatment will be scheduled after patients' first period.
  Interventions: Procedure: LLETZ

INTERVENTIONS:
Drug: Aldara 5% Topical Cream — 5% Imiquimod cream (1 sachet) will be administered via menstrual cup, before going to sleep, 3 times per week for 16 weeks. Menstrual cup will be inserted in the vagina for a duration of 6-8 hours. In case of severe side effects applications can be reduced to twice per week and if side effects are persistent, to once per week. For maximum control of cervical disease, control colposcopy with a PAP smear and a punch biopsy will be scheduled at 10 weeks to rule out progression, and at 20 weeks after treatment initiation to evaluate treatment success. At 20 weeks, biopsies will be performed at the locations where lesions were previously present, and if there are any new lesions present, additional biopsies will be performed. In case of disease progression or persistence, treatment with LLETZ will be offered.
  Other Names: Zyclara, imiquimod
  Arms: Treatment with imiquimod
Procedure: LLETZ — LLETZ will be performed in an outpatient setting with local anesthesia, using KLS Martin Maxium with loop devices ranging from 10 mm to 20 mm in size. The excision will be performed using monopolar current with a cut frequency set to 100-150 W. Treatment success will be evaluated in accordance with our national guidelines 24 weeks after the procedure using a PAP smear with or without a punch biopsy.
  Other Names: LEEP
  Arms: Treatment with LLETZ

SUMMARY:
Purpose: There are limited data on the success of conservative treatment of high-grade cervical squamous intraepithelial lesions (HSIL) with imiquimod directly compared to standard of treatment with LLETZ. LLETZ as standard treatment is possibly associated with premature labour, higher subfertility rate and a higher rate of spontaneous abortion. Since premature delivery is one of the most important causes of perinatal morbidity and mortality, alternative conservative methods for SIL treatment are constantly being evaluated. The immunomodulator imiquimod is one of the main target compounds for treating HSIL.

Primary objective: to establish the efficacy of treatment with imiquimod (experimental arm) and compare it to the standard treatment with LLETZ (control arm).

Secondary objective:

* incidence and severity of the side effects in both groups;
* need for treatment with LLETZ two years after primary treatment with imiquimod in the experimental arm or re-treatment with LLETZ two years after primary treatment with LLETZ in the control arm;
* modulatory effect of imiquimod on immunoregulatory molecules.

Study design: Single-centre randomized controlled intervention trial.

Study population: 104 women with HSIL (52 in each arm).

Intervention:

- randomization in two arms:

1. Experimental arm (imiquimod): treatment for 16 weeks with 5% imiquimod.
2. Control arm (LLETZ).

Successful treatment in the experimental arm is defined as absence of histological HSIL in diagnostic biopsies at 20-week follow-up (4 weeks after treatment completion) and in the control arm successful treatment is defined as absence of cytological HSIL in cytology 6 months after LLETZ (same as in our national guidelines).

DETAILED DESCRIPTION:
Imiquimod is one of the target topical drugs for treating HSIL. It is a Toll-like receptor 7 agonist that acts locally so that it induces cellular response, which can aid in the regression of HPV-associated lesions. Imiquimod is currently used for treating genital warts. In vitro studies have shown promising effects in the treatment of several diseases, such as endometrial, cervical and prostate cancer, endometriosis, melanoma, and cervical and vulvar intraepithelial lesions. Clinical studies are however lacking. With this in mind, the aim of our study was to evaluate whether topical treatment of HSIL with imiquimod is comparable to standard treatment with LLETZ. As mentioned in the Brief summary, we have set different outcome measures in the experimental and control arm. The different outcome measures were based on moderate accuracy of PAP smear, therefore in order to minimize potential progression of cervical disease to cancer and to avoid LLETZ and possible overtreatment and to assess as accurately as possible the potential residual disease, colposcopy with biopsies will be performed 4 weeks after treatment with imiquimod is completed (20th week after treatment initiation). Follow up after LLETZ will performed using cytology (PAP smear), which is in concordance with our national guidelines. Biopsies will be performed in case of clinically visible lesions. Secondary outcomes of the study are the incidence and severity of the side effects in both groups, which will be evaluated during and after treatment using the 5th version of the Common Terminology Criteria for Adverse Events (CTCAE) guidelines. Other secondary outcomes, namely the need for treatment with LLETZ two years after primary treatment with imiquimod in the experimental arm or re-treatment with LLETZ two years after primary treatment with LLETZ in the control arm, respectively, and the modulatory effect of imiquimod on immunoregulatory molecules are expected to be available in three years' time after treatment is completed in all patients in both arms.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed and previously untreated HSIL in women aged 18 to 35 years or up to 40 years in case of nulliparity;
* satisfactory colposcopy (i.e., fully visible lesion and transformation zone);
* negative pregnancy test;
* safe contraception;
* signed, informed consent.

Exclusion Criteria:

* previously diagnosed HSIL or AIS;
* previous LLETZ or classical conisation;
* concomitant vulvar or vaginal lesion or neoplasia;
* other malignancies;
* insufficient colposcopy;
* pregnancy or lactation;
* known hypersensitivity to imiquimod;
* any known contraindications to immunotherapy;
* known HIV or acute or chronic hepatitis;
* immune deficiency;
* participation in any other ongoing clinical trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy of 5% imiquimod cream for treatment of HSIL compared to standard treatment with LLETZ defined as absence of HSIL in both arms (histological in experimental arm and cytological in control arm). | 20 weeks after treatment initiation in experimental arm and 6 months after LLETZ in control arm.
  Defined as following:
  * for experimental (imiquimod) treatment arm: absence of histological HSIL (CIN1 or less) in diagnostic biopsies at colposcopy at 20 weeks;
  * for control (LLETZ) arm: absence of cytological HSIL at 6 months follow-up.

SECONDARY OUTCOMES:
Prevalence and severity of the side effects in both arms. | 10 weeks and 20 weeks after treatment initiation in experimental arm and 20 weeks after LLETZ in control arm.
  Incidence and severity of side effects scored by the 5th version of the Common Terminology Criteria for Adverse Events (CTCAE) guidelines.
Need for LLETZ or repeated LLETZ following primary treatment. | 2 years after primary treatment.
  The need for treatment with LLETZ two years after primary treatment with imiquimod in the experimental arm or re-treatment with LLETZ two years after primary treatment with LLETZ in the control arm
Immunoregulatory effect of imiquimod. | 2 years after primary treatment.
  Modulatory effect of imiquimod on immunoregulatory molecules.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

REFERENCES:
- [Background] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Background] de Witte CJ, van de Sande AJ, van Beekhuizen HJ, Koeneman MM, Kruse AJ, Gerestein CG. Imiquimod in cervical, vaginal and vulvar intraepithelial neoplasia: a review. Gynecol Oncol. 2015 Nov;139(2):377-84. doi: 10.1016/j.ygyno.2015.08.018. Epub 2015 Aug 31. PMID 26335596
- [Background] Koeneman MM, Kruse AJ, Kooreman LFS, Zur Hausen A, Hopman AHN, Sep SJS, Van Gorp T, Slangen BFM, van Beekhuizen HJ, van de Sande M, Gerestein CG, Nijman HW, Kruitwagen RFPM. TOPical Imiquimod treatment of high-grade Cervical intraepithelial neoplasia (TOPIC trial): study protocol for a randomized controlled trial. BMC Cancer. 2016 Feb 20;16:132. doi: 10.1186/s12885-016-2187-3. PMID 26897518
- [Background] Jancar N, Mihevc Ponikvar B, Tomsic S. Cold-knife conisation and large loop excision of transformation zone significantly increase the risk for spontaneous preterm birth: a population-based cohort study. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:245-9. doi: 10.1016/j.ejogrb.2016.06.005. Epub 2016 Jun 20. PMID 27359080
- [Derived] Cokan A, da Silva NCH, Kavalar R, But I, Pakiz M, Andrade de Oliveira S, Dos Santos Gomes FO, da Silva RS, Peixoto CA, Lucena-Silva N. Modulation of sHLA-G, PD-1, and PD-L1 Expression in Cervical Lesions Following Imiquimod Treatment and Its Association with Treatment Success. Cancers (Basel). 2024 Mar 25;16(7):1272. doi: 10.3390/cancers16071272. PMID 38610950